CLINICAL TRIAL: NCT07054645
Title: Evaluation of the Effects of Elderberry-Based Anthocyanin-Enriched Functional Chewing Gum on Cognitive Functions and Oral Microbiota in Older Adults: A Double-Blind, Randomized Controlled Trial
Brief Title: Elderberry Functional Gum and Cognitive & Oral Health in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Gul Akduman, Dr., Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MAKU-AKDUMAN-1002-2025
Record Dates: First submitted 2025-06-19; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment (MCI); Aging; Oral Microbiome
Keywords: Elderberry; Anthocyanins; Chewing Gum; Functional Food; Transmucosal Delivery; Oral Microbiota; Cognitive Function; MoCA; Aging; Mild Cognitive Impairment; Geriatric Nutrition; Randomized Controlled Trial
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group design. Participants are randomly assigned to either the intervention group (elderberry-based anthocyanin chewing gum) or the placebo group. Both groups are assessed at baseline and after 6 weeks of intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomly assigned to intervention or placebo groups using computer-generated permuted block randomization (block size = 4). Allocation sequences will be created by an independent researcher. Gums will be packaged in identical blister packs labeled with alphanumeric codes that do not reveal group assignment. Only the randomization coordinator will have access to the allocation key. Investigators and outcome assessors will be blinded throughout the study. Cognitive tests and saliva sampling will be conducted by trained staff unaware of group assignment, under standardized conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elderberry Chewing Gum Group (Experimental): Participants receive chewing gum containing standardized elderberry anthocyanins twice daily for 6 weeks
  Interventions: Dietary Supplement: Elderberry Anthocyanin Chewing Gum
- Placebo Arm Title (Placebo Comparator): Participants receive anthocyanin-free chewing gum matched in appearance and taste, twice daily for 6 weeks
  Interventions: Dietary Supplement: Placebo Chewing Gum

INTERVENTIONS:
Dietary Supplement: Elderberry Anthocyanin Chewing Gum — Participants receive a functional chewing gum containing encapsulated elderberry (Sambucus nigra L.) anthocyanins standardized for cyanidin-3-glucoside and cyanidin-3-sambubioside. The gum is formulated to be geriatric-friendly (soft, low-elasticity) and is administered twice daily for 6 weeks. It enables transmucosal polyphenol delivery through buccal absorption.
  Arms: Elderberry Chewing Gum Group
Dietary Supplement: Placebo Chewing Gum — Participants receive a placebo chewing gum identical in appearance, taste, and texture to the active gum but containing no elderberry anthocyanins or bioactive compounds. The gum is administered twice daily for 6 weeks to match the intervention group.
  Arms: Placebo Arm Title

SUMMARY:
Globally, the aging population is increasing rapidly, leading to a dramatic rise in the prevalence of Alzheimer's disease and other types of dementia. Neurodegenerative disorders are characterized by pathological hallmarks such as β-amyloid (Aβ) plaque accumulation, tau protein aggregation, synaptic loss, and widespread neuroinflammation. These processes impair key cognitive domains including attention, memory, executive function, and orientation, hindering independent daily functioning.

Beyond cognitive decline, neurodegenerative diseases are associated with a marked deterioration in oromotor functions, such as chewing and swallowing. Mastication plays a critical role not only in digestion but also in neuro-sensory stimulation. Trigeminal nerve signaling activated by chewing enhances neurotransmitter release, boosts neurotrophic factor production (e.g., BDNF), and facilitates Aβ clearance, thereby supporting synaptic plasticity and reducing inflammation. Neuroimaging studies have shown that a higher number of functional occlusal pairs is associated with increased gray and white matter volume in regions affected early in Alzheimer's disease.

Systematic reviews have identified poor mastication and tooth loss as risk factors for cognitive decline and dementia. Mechanistically, loss of afferent input from the oral cavity-due to tooth loss, reduced chewing force, prosthetic use, or muscle atrophy-leads to reduced brain stimulation, diminished neurotrophic support, and impaired cerebral blood flow. Thus, geriatric-friendly chewing gum formulations with low elasticity and ease of chewing have been recommended.

Chewing gum is a promising vehicle for functional compounds due to its potential for transmucosal absorption and cognitive stimulation. Randomized controlled trials have shown that both active and inactive gums improve attention and reduce error rates in cognitive tasks, highlighting the beneficial effects of mastication.

Another emerging target for cognitive enhancement is the oral microbiota, a complex ecosystem of over 700 bacterial species. Dysbiosis in this ecosystem has been linked to neurological outcomes via inflammatory and neurotoxic pathways. Certain pathogens, such as Porphyromonas gingivalis, have been detected in the brains of Alzheimer's patients. Moreover, metagenomic studies have shown that reduced salivary microbial diversity correlates with poorer cognitive performance, even in young adults.

Elderberry (Sambucus nigra L.) is rich in anthocyanins (e.g., cyanidin-3-glucoside, cyanidin-3-sambubioside) with strong antioxidant and anti-inflammatory properties. Literature shows that polyphenols can be absorbed via buccal and sublingual mucosa, bypassing first-pass metabolism and providing faster systemic effects. However, the impact of anthocyanin-enriched chewing gum on oral microbiota and cognitive function has not yet been systematically investigated.

This study aims to develop and evaluate a geriatric-friendly functional chewing gum enriched with standardized elderberry anthocyanins. The intervention targets dual mechanisms-neurophysiological and microbial-to support cognitive health and balance oral microbiota in older adults.

DETAILED DESCRIPTION:
This study is a double-blind, randomized controlled clinical trial designed to evaluate the impact of an elderberry-based functional chewing gum on cognitive function and oral microbiota in older adults.

The chewing gum intervention contains encapsulated anthocyanins derived from Sambucus nigra L., standardized for cyanidin-3-glucoside and cyanidin-3-sambubioside content, and formulated specifically for elderly individuals. The gum is designed to be soft-textured, low in elasticity, and easy to chew. It also allows transmucosal absorption through buccal and sublingual pathways, offering a rapid delivery system for polyphenols.

The study will enroll 34 participants aged 60 and above, with mild cognitive impairment (MoCA 20-25), divided equally into intervention and placebo groups. Participants will chew one gum twice daily for 6 weeks. During the intervention, participants will follow a berry-free diet to eliminate potential confounding sources of polyphenols.

Pre- and post-intervention assessments will include:

* Cognitive performance using MoCA and Stroop Color-Word Test (TBAG form)
* Salivary analysis for flow rate, pH, antioxidant capacity (FRAP), and total phenolic content (Folin-Ciocalteu)
* Microbiota profiling via 16S rRNA sequencing (in a subsample) and culturing of S. mutans and Lactobacillus spp.
* Compliance tracking via daily chewing logs and weekly monitoring

The primary hypothesis is that the anthocyanin-enriched gum will:

* Enhance cognitive performance,
* Improve oral microbial diversity,
* Reduce cariogenic bacteria (e.g., S. mutans),
* Increase salivary antioxidant capacity. Secondary goals include evaluating the gum's acceptability using a 9-point hedonic scale and assessing the stability of anthocyanin content over time.

Anthocyanin content and release will be validated by HPLC and pH-differential spectrophotometry, and stability will be tested over a 6-month period according to ICH guidelines. Statistical analysis will be performed using ANOVA, t-tests, and linear models adjusting for education and age.

This multidisciplinary study integrates dietary polyphenols, oral delivery systems, salivary biomarkers, microbiome science, and cognitive neuroscience in a novel, geriatric-focused intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 60 and over
* Individuals with mildly reduced cognitive function using the MoCA test (MoCA score: 20-25)
* Those with stable systemic diseases (e.g. HT, controlled DM)
* Those with adequate dental health (≥20 natural teeth or no chewing problems with functional prosthesis)
* Non-smokers and those who use regular medication and do not use antibiotics or antiseptic mouthwashes that could seriously affect the oral microbiota
* Individuals who are willing to participate in the study and can give written consent

Exclusion Criteria:

* Moderate to severe dementia (MoCA < 20)
* Presence of active infection or systemic inflammatory disease
* Temporomandibular joint disorders affecting gum chewing function
* Use of probiotics, prebiotics, or antibiotics within the last three months
* Known allergy to elderberry or its components

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive Function Assessed by MoCA (Montreal Cognitive Assessment) Score | Baseline and Week 6
  The MoCA score (0-30) will be used to assess global cognitive function. A higher score indicates better cognitive performance. Measurements will be taken at baseline and at 6 weeks.

SECONDARY OUTCOMES:
Change in Executive Function Assessed by Stroop Test | Baseline and Week 6
  Cognitive flexibility and executive control will be assessed using the Stroop Color-Word Test (TBAG form). The interference score (difference in reaction time between incongruent and color conditions) will be used as the main outcome. Unit of Measure: milliseconds (ms)
Change in Alpha Diversity Assessed by Shannon Index | Baseline and Week 6
  lpha diversity of oral microbiota will be assessed using the Shannon Index, based on 16S rRNA gene sequencing. Unit of Measure: Shannon diversity index (unitless)
Change in Beta Diversity Assessed by UniFrac and Bray-Curtis Distances | Baseline and Week 6
  Beta diversity of oral microbiota will be assessed using UniFrac and Bray-Curtis distances, based on 16S rRNA gene sequencing. Unit of Measure: Distance metric (unitless)
Change in Salivary Flow Rate | Baseline and Week 6
  Unstimulated whole saliva will be collected for 5 minutes. Flow rate will be calculated and expressed in mL/min. Differences from baseline to week 6 will be analyzed.
Change in Salivary pH | Baseline and Week 6
  Salivary pH will be measured from unstimulated whole saliva samples collected over 5 minutes. Differences from baseline to week 6 will be analyzed.Unit of Measure: pH value (unitless)
Change in Salivary Total Antioxidant Capacity (FRAP Method) | Baseline and Week 6
  The Ferric Reducing Antioxidant Power (FRAP) assay will be used to evaluate the total antioxidant capacity of unstimulated saliva samples. Results will be expressed as micromoles of Fe²⁺ equivalents per milliliter (µmol Fe²⁺/mL).
Change in Salivary Total Phenolic Content (Folin-Ciocalteu Method) | Baseline and Week 6
  The Folin-Ciocalteu colorimetric method will be used to quantify the total phenolic content in unstimulated saliva. Results will be reported as milligrams of gallic acid equivalents per milliliter (mg GAE/mL).
Change in Salivary Streptococcus mutans Count | Baseline and Week 6
  Salivary concentration of Streptococcus mutans will be assessed using microbiological culturing on selective agar. Results will be reported as colony-forming units per milliliter (CFU/mL).
Change in Salivary Lactobacillus spp. Count | Baseline and Week 6
  Salivary concentration of Lactobacillus spp. will be assessed using microbiological culturing on selective agar. Results will be reported as colony-forming units per milliliter (CFU/mL).
Product Acceptability Score (Hedonic Scale) | Initial Exposure and Week 6
  Participants will evaluate the taste, texture, aroma, and overall liking of the chewing gum using a 9-point hedonic scale (1 = Dislike extremely, 9 = Like extremely). Higher scores indicate greater acceptability.
  Unit of Measure: Score (1-9)

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Akif Ersoy University, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and privacy concerns. The study protocol did not include participant consent for open data sharing, and the dataset contains potentially identifiable health information.